CLINICAL TRIAL: NCT05166226
Title: The Reliability and Validity of the PortionSize™ and MyFitnessPal Apps (Study 2: Semi-controlled, Free-living Evaluation)
Brief Title: PortionSize Study 2 Free-Living Evaluation
Status: Active, not recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, PBRC Professor, Director - Ingestive Behavior Laboratory, Pennington Biomedical Research Center
Other Study IDs: PBRC 2019-061
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Dietary Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective is to test the accuracy of the PortionSize™ app and the MyFitnessPal© app at measuring energy and nutrient intake in free-living conditions. Participants will use PortionSize™ and MyFitnessPal apps in separate periods to test the accuracy of the respective apps.

DETAILED DESCRIPTION:
Accurately quantifying food intake is vital to promoting health and reducing chronic disease risk. Food intake encompasses energy intake, nutrient intake (macronutrients, micronutrients, vitamins, minerals), and intake of various food groups (e.g., fruits, vegetables), and thus reflects the nutritional status of individuals. Nutrition affects disease risk, including risk of developing obesity, diabetes, and cancer, all of which negatively affect the United States (U.S). Nonetheless, accurate assessment of food and nutrient intake has remained challenging, despite an improvement in methods. Self report methods, namely food records, are a mainstay of nutritional epidemiology research, with food recall being another popular method. These methods rely on the participant to accurately estimate portion size and, for food recall, remember what was consumed. The accuracy of these methods have been questioned and the problems with human recall have been comprehensively outlined. As a result, there remains a significant need for methods that are sufficiently accurate to provide researchers with good outcome data and to guide health promotion efforts.

The PortionSize™ app was designed by our laboratory to overcome the limitations outlined above, and to guide users to follow specific diets. PortionSize™ relies on users capturing images of their food selection and waste. Food intake data are immediately provided since the user relies on built in tools, including templates, to estimate portion size. However, despite promising early indications, the PortionSize™ app has yet to be fully validated. Determining the accuracy and reliability of PortionSize™ is vital before the app can be used by people to obtain immediate feedback about their food intake. We accordingly aim to test the reliability and validity of PortionSize™ in a semi-controlled free-living environment using food provision, where participants consume pre-weighed food from a cooler and return the plate waste in the cooler. We will also test the reliability and validity of the MyFitnessPal app in the same semi-controlled free-living environment. The accuracy of the apps will also be compared to each other.

ELIGIBILITY:
Inclusion Criteria:

Male or female, age 18-62 years

* Body mass index (BMI) 18.5-50 kg/m2
* Subjects who are capable of giving informed consent and complying with all study procedures/requirements.
* Ownership of an iPhone model 6s or later, which the participant is willing to use for the study
* Access to Apple ID, password, and email address and willing to use them during the study
* Willing to use data and any accompanying charges as part of study participation
* Willing to complete all study procedures and adhere to study visit timelines
* Willing to be re-contacted for future research and/or follow-up

Exclusion Criteria:

* Active cancer diagnosis (excluding some melanomas)
* Have been 6-month weight unstable (gain/loss >10 lbs in last 6 months)
* Undergoing weight loss treatment
* PBRC employee, as previous reviewers argued that they are not representative of the community
* Women who are currently pregnant or breastfeeding (self-reported)
* Diagnosed with an uncontrolled thyroid disorder (controlled = 3 months of medication)
* Have had or plan to have weight loss surgery (gastric band removal may be allowed at PI discretion)
* Allergic to or unwilling to eat study foods provided (exceptions made at the discretion of the PI)
* Consume >28 alcoholic beverages per week
* Anyone severely immunocompromised
* Any condition or circumstance that in the judgement of the PI could interfere with study participation

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants ages 18 to 62 in the Baton Rouge, LA area
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Corby K Martin, PhD, Principal Investigator — Pennington Biomedical Research Center; John W Apolzan, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Diktas HE, Lozano CP, Saha S, Broyles ST, Martin CK, Apolzan JW. Validity of the PortionSize and MyFitnessPal Smartphone Applications for Estimating Dietary Intake: A Randomized Crossover Clinical Trial. J Nutr. 2025 Dec;155(12):4296-4306. doi: 10.1016/j.tjnut.2025.09.027. Epub 2025 Sep 27. PMID 41022156

RESULTS

PARTICIPANT FLOW:
Groups:
- PortionSize Followed by MyFitnessPal: This was a within-subjects, randomized, counterbalanced crossover design. Each participant completed two testing periods: Period 1 and Period 2. Participants were randomly assigned to one of two sequences: (1) PortionSize followed by MyFitnessPal, or (2) MyFitnessPal followed by PortionSize. PortionSize followed by MyFitnessPal group used the PortionSize app to estimate dietary intake during the first study period and switched to MyFitnessPal for the second period.
- MyFitnessPal Followed by PortionSize: This was a within-subjects, randomized, counterbalanced crossover design. Each participant completed two testing periods: Period 1 and Period 2. Participants were randomly assigned to one of two sequences: (1) PortionSize followed by MyFitnessPal, or (2) MyFitnessPal followed by PortionSize. MyFitnessPal followed by PortionSize group used the MyFitnessPal app to estimate dietary intake during the first study period and switched to PortionSize for the second period.
Period: Overall Study
Arm/Group | PortionSize Followed by MyFitnessPal | MyFitnessPal Followed by PortionSize
Started | 23 | 22
Completed | 23 | 21
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All 44 participants that completed the study
Arm/Group | All Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 44
BMI [Mean (Standard Deviation); unit: kilograms per square meter (kg/m²)] | 28.6 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Energy (Kilocalorie or kcal) Intake
Description: The primary analyses assessing equivalence between PortionSize™ and the criterion measure (and MyFitnessPal and the criterion measures) will rely on equivalence testing using the Two One-side T-test (TOST) method. The null hypothesis of an equivalence tests is that the means are nonequivalent, i.e., the confidence interval of the mean of the test condition exceeds the pre-specified error bound. The alternative hypothesis is that the means are equivalent, and the mean difference between the experimental method and gold standard is hypothesized to be zero. Differences in error from PortionSize™ compared to error from MyFitnessPal will be assessed using dependent samples t-tests, with error calculated as the difference between each experimental method and the criterion variable (e.g., energy intake values from PortionSize™ minus energy intake values from weighed foods). These procedures will also produce results indicating if the error from each method differs from zero.
Time Frame: Mean daily energy intake averaged across 3 day free-living period of each PortionSize app and MyFitnessPal app intervention.
Population: All participants completed two study periods using both the PortionSize and MyFitnessPal apps. Outcome measures are summarized by intervention (PortionSize vs. MyFitnessPal), pooling data across all participants regardless of the order in which apps were used.
Measure: Mean (Standard Deviation); unit: kcal/day
Groups:
- PortionSize: This was a within-subjects, randomized, counterbalanced crossover design. Each participant completed two testing periods: Period 1 and Period 2. Participants were randomly assigned to one of two sequences of interventions: (1) PortionSize followed by MyFitnessPal, or (2) MyFitnessPal followed by PortionSize.
- MyFitnessPal: This was a within-subjects, randomized, counterbalanced crossover design. Each participant completed two testing periods: Period 1 and Period 2. Participants were randomly assigned to one of two sequences: (1) PortionSize followed by MyFitnessPal, or (2) MyFitnessPal followed by PortionSize.
Arm/Group | PortionSize | MyFitnessPal
Number analyzed (Participants) | 44 | 44
kcal/day | 2128.8 (762.1) | 2120.0 (650.1)

ADVERSE EVENTS:
Time Frame: 3 days in free-living conditions per intervention
Groups:
- PortionSize: Participants completed three days using the PortionSize app during one of the two study periods. Adverse events are reported for all participants during this intervention period, regardless of sequence.
- MyFitnessPal: Participants completed three days using the MyFitnessPal app during one of the two study periods. Adverse events are reported for all participants during this intervention period, regardless of sequence.
Arm/Group | PortionSize | MyFitnessPal
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT05166226/Prot_SAP_000.pdf